CLINICAL TRIAL: NCT00544505
Title: Pre-operative Chemotherapy in Operable Breast Cancer, Phase III Study Comparing a Short Intensive Pre-operative Chemotherapy With the Same Therapy Initiated Shortly After Surgery(Peri-operatively)(POCOB)EORTC 10902)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#931-006
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; EC regimen

INTERVENTIONS:
Drug: Fluorouracil/Epirubicin/Cyclophosphamide — Phase III Comparison of Preoperative vs Postoperative FEC (Fluorouracil/Epirubicin/Cyclophosphamide) in Women with Operable Breast Cancer

SUMMARY:
Pre-operative chemotherapy in operable breast cancer, phase III study comparing a short intensive pre-operative chemotherapy with the same therapy initiated shortly after surgery (peri-operatively) (POCOB) (EORTC 10902)

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

* Palpable, operable breast cancer that has been diagnosed by core needle biopsy (mandatory for T1c tumors) or fine needle aspiration within 21 days prior to entry
* Stage T1c-4b, N0-1, M0

Hormone receptor status:

* Not specified
* No bilateral breast cancer

Prior/Concurrent Therapy:

* No previous treatment for breast cancer

Biologic therapy:

* Not specified

Chemotherapy:

* No previous chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Core needle biopsy or fine needle aspiration within 21 days prior to entry
* Repeated core needle biopsy permitted

Patient Characteristics:

Age:

* 16 to 70

Sex:

* Women only

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Hematopoietic:

* WBC at least 4,000
* Platelets at least 100,000

Hepatic:

* Bilirubin no greater than 2.8 mg/dL (50 micromoles/L)

Renal:

* Creatinine no greater than 1.3 mg/dL (120 micromoles/L)

Cardiovascular:

* No congestive heart failure
* No significant arrhythmia
* No bilateral bundle branch block
* No recent myocardial infarction
* No uncontrolled hypertension (diastolic pressure greater than 110 mm Hg)

Other:

* No male breast cancer
* No pregnant or nursing women
* No second malignancy except adequately treated:

  * Nonmelanomatous skin cancer
  * Cervical cancer

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy | overall

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Ezzat, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia